CLINICAL TRIAL: NCT05990439
Title: Baby-Feed Web Application for Infant Caregivers to Improve Diets and Weight Gain
Acronym: BabyFeed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Academy of Nutrition and Dietetics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 23-0409
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Investigator
Masking Description: randomization, assignment of arms, assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm will have full access to the Baby-Feed web application. It was based on the Social Cognitive Theory and the Health Self-Empowerment Theory.
  It provides automatic feedback based on the infant FFQ, showing the total amounts of each food group consumed (milk, protein foods, whole and refined grains, fruits, vegetables, juices, sugary beverages, sweets, and salty snacks) with automated feedback of which are consumed adequately or above/below the recommendations.
  * Recommendations: this section displays the amount recommended for each food group by age group.
  * Tracking: This is a short form that asks participants to evaluate if they gave the recommended amounts of each food group in the past week.
  * Weight gain tracker: parents are asked to input the weight and length of their baby and it shows graphically how the baby is progressing.
  Interventions: Behavioral: Baby-Feed
- Control group (Placebo Comparator): Participants randomized to the control arm (n=80) will have limited access to certain components of the Baby-Feed web application, such as the online infant FFQ to complete it at the same intervals (before the 4-month, 6-month, and 9-month well-child visits) and infant's weight and length as recorded in the well-child visits, but without any automatic results or feedback. The control group will have a separate user access to the Baby-Feed web application that only allows them to complete the required information without being able to see results, feedback, tracking, recommendations, or resources.
  Interventions: Behavioral: Limited access to the Baby-Feed web application

INTERVENTIONS:
Behavioral: Baby-Feed — The Baby-Feed web application was developed by the researchers of this application at Florida International University. It was designed based on a validated infant food frequency questionnaire (FFQ) developed by our group. The Social Cognitive Theory (SCT) and the Health Self-Empowerment Theory (HSET) were used in the development of the different components. The main intervention component is showing automatic results on how well parents are feeding their infants, upon completion of the infant FFQ, showing results on which food groups are consumed at the recommended level, which are consumed above and which are consumed below. It also shows a growth chart showing how the baby is progressing when they add their baby's weight and length. The website also includes a tracking system with short questions asking about their weekly progress and the recommendations to review frequently, if needed.
  Arms: Intervention
Behavioral: Limited access to the Baby-Feed web application — Limited access to the Baby-Feed web application, with only the options of completing the FFQ and inputing their baby's weight and length.
  Arms: Control group

SUMMARY:
This study will test the Baby-Feed web platform among 160 parents with infants aged 1-3 months at the time of enrollment and follow them through their 9-month well-child visit (about a total of 6 months) using a mixed-methods approach (randomized control trial with qualitative interviews).

DETAILED DESCRIPTION:
This study will test the Baby-Feed web platform among 160 parents with infants aged 1-3 months at the time of enrollment and follow them through their 9-month well-child visit (about a total of 6 months) using a mixed-methods approach (randomized control trial with qualitative interviews). This age range was chosen as this is the period in which parents initiate and continue complementary foods in their infants' diets. Procedures: Participants randomized to the intervention arm (n=80) will have full access to the Baby-Feed web application and receive automated weekly text messages to complement the information received in Baby-Feed and to remind them to access the web application. Within the Baby-Feed platform, the intervention arm will assess the online infant FFQ to complete it at the required intervals (before the 4-month, 6-month, and 9-month well-child visits) and receive automatic feedback for obtaining recommended intake of food groups as well as input bi-weekly tracking goals. They will also record their infant's weight and length as provided from the well-child visits, which will plot on the WHO CDC 0-24 months growth chart and provide feedback to their infant's growth pattern. Caregivers will also have access to educational resources to aid them in reading and viewing appropriate infant guidance. Participants randomized to the control arm (n=80) will have access to certain components of the Baby-Feed web application, such as the online infant FFQ to complete it at the same intervals (before the 4-month, 6-month, and 9-month well-child visits) and infant's weight and length as recorded in the well-child visits, but without any automatic results or feedback. Risks and anticipated benefits: It is anticipated that this trial will have minimal risks as it is self-reported data only. Anticipated benefits include caregivers receiving dietary and weight gain guidance during the study which may assist with optimal nutritional and weight status. The importance of the knowledge that may reasonably be expected to result: The importance of this knowledge could lead to public use of the Baby-Feed web application leads to improvements in diet and weight gain during this critical time of growth and by potentially becoming a routine and accessible tool for clinicians to recommend their patients to support optimal growth and development for infants

ELIGIBILITY:
Inclusion Criteria:

* 1-3 months old at time of enrollment, term healthy infant, any weight status, parent/family member must be primary caretakers, have internet access, agree to receive text messaging service for communication and reminders, willing to participate for full study duration, and English or Spanish language literate.

Exclusion Criteria:

* Infants with special diets, preterm birth (<37 weeks), caregiver inability to consent to participate, unwillingness to be randomized, and unable to read in English or Spanish.

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 155 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Diet Quality | 9 months
  It will be analyzed from the responses to the infant FFQ using the Diet Quality Index Score (DQIS)
Rate of weight gain | 9 months
  It will be analyzed from the plotted weight and length as recorded by caregivers in the WHO gender-specific growth chart table in Baby-Feed after each well-child visit (4, 6, and 9 months) to calculate weight-for-length z-score.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Palacios, PhD, Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided